CLINICAL TRIAL: NCT05302635
Title: The Effect of Simulation-based Training in Nasogastric Tube Application in Children on the Clinical Skills of Nursing Students: An Experimental Study
Brief Title: The Effect of Simulation-based Training on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Mujde CALIKUSU Incekar, Assistant Professor, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YIU-M-CI-002
Record Dates: First submitted 2022-02-13; First posted 2022-03-31 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Simulation; Education; Learning; Clinical Skills; Child
Keywords: Simulation; Nursing student; Clinical skills; Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated group (Experimental): Students will be given training on nasogastic tube insertion and practice will be demonstrated in the laboratory based on the demonstration method and checklists, and will continue until students learn. Forms will be applied to students as a pre-test. A pilot scenario will be applied to two volunteer fourth year students.
  Prebriefing: Students will be informed. Students will implement the scenario in the simulation laboratory and will wear uniforms. The student will be given 5 minutes for preparation, the application will be taken one by one and 15 minutes will be given for practice. Researchers will only observe during this time. During the application, the student will be scored according to the checklist. Students will be recorded with video.
  Debriefing: Immediately after the end of the scenario, a debriefing session will be held with groups of 5 people. Feedback will be given on students' performance. Each session will last 20-30 minutes. Students will be given a post-test.
  Interventions: Other: Simulated group
- Control group (No Intervention): Students will be given training on nasogastric tube insertion and nasogastric tube application will be demonstrated with the demonstration method in the laboratory and will continue until students learn. Forms will be applied to students as a pre-test. A pilot scenario will be applied to two volunteer fourth year students.
  Prebriefing: Students will be informed. Students will apply the scenario on the model in the skill laboratory and will wear uniforms. The student will be given 5 minutes for preparation. Students will be taken to the application one by one and 15 minutes of practice time will be given. During the application, the student will be scored according to the checklist. Students will be recorded with video.
  Debriefing: Immediately after the end of the scenario, a debriefing session will be held with groups of 5 people. Feedback will be given on students' performance in the debriefing session. Each session will last 20-30 minutes. Students will be given a post-test.

INTERVENTIONS:
Other: Simulated group — Students will be given training on nasogastic tube insertion and practice will be demonstrated in the laboratory based on the demonstration method and checklists, and will continue until students learn. Forms will be applied to students as a pre-test. A pilot scenario will be applied to two volunteer fourth year students.
  Prebriefing: Students will be informed. Students will implement the scenario in the simulation laboratory and will wear uniforms. The student will be given 5 minutes for preparation, the application will be taken one by one and 15 minutes will be given for practice. Researchers will only observe during this time. During the application, the student will be scored according to the checklist. Students will be recorded with video.
  Debriefing: Immediately after the end of the scenario, a debriefing session will be held with groups of 5 people. Feedback will be given on students' performance. Each session will last 20-30 minutes. Students will be given a post-test.
  Arms: Simulated group

SUMMARY:
This research will be carried out with the aim of making this practice practical with simulation-based training and improving cognitive, affective and psychomotor skills, and then applying it in the clinic, before applying the nasogastric tube placement application, which is included in enteral nutrition, to the child in the clinic.

DETAILED DESCRIPTION:
The fact that children react according to their age and cannot be considered separately from their families makes it difficult for nurse students to apply to the child group. When it comes to interventions that may cause stress/pain/discomfort, it can be even more difficult to manage the reactions of the child and family. By using the simulation method, the problems that make this type of teaching difficult can be reduced.For this reason, the aim of this study is for student nurses to make this practice practical with simulation-based training and to develop cognitive, affective and psychomotor skills before applying nasogastric tube placement, which is included in enteral nutrition, to a real child in the clinic, and then to apply it in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Studying in the 3rd year of the Faculty of Health Sciences, Nursing Department of Yüksek İhtisas University and Biruni University,
* Having successfully completed the clinical application of the Fundamentals of Nursing course, Internal Medicine Nursing course and Surgical Diseases Nursing course and not repeating the grade,
* Those who will take the Child Health and Diseases Nursing course for the first time,
* Students who volunteer to participate in the research will be included.

Exclusion Criteria:

* Having received training on enteral nutrition in children,
* Simulation training,
* Students coming from other health departments (such as anaesthesia, laboratory technician, elderly health personnel) or from health vocational high schools as nursing will be excluded.
* Students who want to exit the research at any stage of the research will be excluded from the research.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy - Competence Scale | immediately after training on nasogastic tube insertion and practice in the laboratory
  The scale was developed by Sherer et al. (1982). The scale, which does not belong to any subjective domain, measures the general perception of self-efficacy - efficacy. The scale consists of 23 items and four subscales. The subscales of the scale are respectively; These are "beginning the behavior", "maintaining the behavior", "Completing the behavior" and "Combating the obstacles". For each item; It is a five-point Likert-type scale as 1 = does not describe me at all, 2 = describes me a little, 3 = is undecided, 4 = describes me well, 5 = describes me very well. A score between 23 and 115 can be obtained from the scale. A high total score from the scale indicates that the individual's self-efficacy-efficacy perception is at a good level. The validity and reliability of the Turkish version of the scale was performed by Gözüm and Aksayan (1999).
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the debriefing session
  The scale was developed by Jeffries and Rizzolo (2006) as 13 items to measure students' simulation activity and self-confidence in learning. Answering the scale for each item; 1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Strongly Agree (Franklin et al., 2014). The Turkish validity and reliability study of the scale was carried out by Unver et al. (2017) and the total number of items decreased to 12.
Clinical Decision Making Scale in Nursing | immediately after training on nasogastic tube insertion and practice in the laboratory
  The Nursing Clinical Decision Making Scale was developed by Jenkins (1983) for nursing students. This scale defines how nursing students perceive clinical decision making based on their own statements. The scale consists of 40 items and four subscales. The subscales of the scale are respectively; These are "Exploring options and ideas", "Exploring goals and values", "Evaluating results", and "Searching for information and adopting new information objectively". Each subscale consists of 10 items. Each item of the scale is evaluated as 5=Always, 4=Often, 3=Sometimes, 2=Rarely, 1=Never. A high score from the scale indicates a high perception of decision making (Jenkins, 1983; Jenkins, 2001). The Turkish validity and reliability of the scale was done by Durmaz Edeer and Sarıkaya (2015).
Nasogastric Tube Placement Checklist | During the application (experimental group= in the simulation laboratory; control group= in the skill laboratory
  The Child Checklist was prepared by the researchers based on the literature (Bindler et al., 2014). The skill performance of the student will be evaluated over a total of 100 points, by scoring each application step according to the degree of importance.

SECONDARY OUTCOMES:
Self-Efficacy - Competence Scale | immediately after the debriefing session
  The scale was developed by Sherer et al. (1982). The scale, which does not belong to any subjective domain, measures the general perception of self-efficacy - efficacy. The scale consists of 23 items and four subscales. The subscales of the scale are respectively; These are "beginning the behavior", "maintaining the behavior", "Completing the behavior" and "Combating the obstacles". For each item; It is a five-point Likert-type scale as 1 = does not describe me at all, 2 = describes me a little, 3 = is undecided, 4 = describes me well, 5 = describes me very well. A score between 23 and 115 can be obtained from the scale. A high total score from the scale indicates that the individual's self-efficacy-efficacy perception is at a good level. The validity and reliability of the Turkish version of the scale was performed by Gözüm and Aksayan (1999).
Clinical Decision Making Scale in Nursing | immediately after the debriefing session
  The Nursing Clinical Decision Making Scale was developed by Jenkins (1983) for nursing students. This scale defines how nursing students perceive clinical decision making based on their own statements. The scale consists of 40 items and four subscales. The subscales of the scale are respectively; These are "Exploring options and ideas", "Exploring goals and values", "Evaluating results", and "Searching for information and adopting new information objectively". Each subscale consists of 10 items. Each item of the scale is evaluated as 5=Always, 4=Often, 3=Sometimes, 2=Rarely, 1=Never. A high score from the scale indicates a high perception of decision making (Jenkins, 1983; Jenkins, 2001). The Turkish validity and reliability of the scale was done by Durmaz Edeer and Sarıkaya (2015).

CONTACTS AND LOCATIONS:
Overall Officials: Sevim SAVAŞER, PhD, Principal Investigator — Biruni University; Hülya ZENGİN, PhD, Principal Investigator — Yuksek Ihtisas University; Gizem KAYA, MsC, Principal Investigator — Biruni University; Bahar ON, MsC, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)